CLINICAL TRIAL: NCT02219438
Title: Continuous Adductor Canal Nerve Blocks: Relative Effects of a Basal Infusion v. Hourly Bolus Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Adductor Canal Basal vs Bolus
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy Human Volunteers
MeSH Terms: interventions — NOP-bolus regimen

STUDY DESIGN:
Intervention Model Description: This is a split-body study in which each study subject receives both treatments: one on each side of the body. Which treatment is applied to which side of the body is randomized (and masked).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only individual aware of the treatment group assignments is the investigational pharmacist who has no interaction with the study subjects. Treatment group assignments were released by the investigational pharmacy only after completion of data collection.
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIGHT side BOLUS and left side basal (Experimental): Bilateral adductor canal catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as hourly bolus doses of 8 mL each a total of 8 times: one at time point zero and 1 on the hour for the following 7 hours. For the left catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 8 hours
  Interventions: Drug: Bolus; Drug: Basal
- RIGHT side BASAL and left side bolus (Active Comparator): Bilateral adductor canal catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 8 hours. For the left catheter, the ropivacaine was administered as hourly bolus doses of 8 mL each a total of 8 times: one at time point zero and 1 on the hour for the following 7 hours.
  Interventions: Drug: Bolus; Drug: Basal

INTERVENTIONS:
Drug: Bolus — An adductor canal catheter was inserted and ropivacaine 0.2% administered as hourly bolus doses of 8 mL each: one at time point zero and then on the hour for 7 additional doses.
  Other Names: hourly bolus doses
Drug: Basal — An adductor canal catheter was inserted and ropivacaine 0.2% administered as a continuous basal infusion (8 mL/h) from time point zero for a total of 8 hours.
  Other Names: continuous basal infusion

SUMMARY:
Patients usually experience moderate-to-severe pain following the knee replacement that is often treated with a femoral nerve block (injection of numbing medicine placed around the main nerve of the knee joint). To make the nerve block last longer, a tiny tube is often placed next to the nerve and numbing medicine is infused for multiple days. However, while the numbing medicine takes away pain, it also decreases sensations, muscle strength, and proprioception (knowing where the leg is in space without looking at it) which greatly increases the risk of falling. Since falling can be catastrophic following major surgery, a femoral nerve blocks are being phased out by surgeons and anesthesiologists. The most-promising replacement is called an adductor canal nerve block. For this new type of block, a perineural catheter is inserted into a small canal in the middle of the upper leg. This canal contains the sensory nerve fibers leading to the knee, and only a single nerve that serves a relatively small muscle. Multiple studies have demonstrated a dramatic increase in muscle strength using the new adductor canal block compared with the traditional femoral block. However, practitioners perceptions of the new block is that it provides insufficient pain control following knee arthroplasty, even though all of the sensory nerves affected with the femoral block are also-theoretically-affected with the adductor canal block. One reason for this difference may be the small canal of the latter which is a relatively tight area in which the numbing medicine might not spread particularly well (due to pressure from surrounding tissues). One way to possibly counter this issue is by providing repeated boluses of the numbing medicine that will improve the medicine's spread relative to a more-traditional slow, continuous ("basal") infusion. This study seeks to compare these two techniques of medication administration through perineural adductor canal catheters:

Our primary aim is to test the hypothesis that, for continuous adductor canal blocks, providing local anesthetic as repeated, hourly bolus doses results in an increased sensory block compared with providing local anesthetic as a continuous basal infusion at an equivalent hourly dose.

As a secondary aim, we hypothesize that, for continuous adductor canal blocks, providing local anesthetic as repeated, hourly bolus doses results in either equivalent or less motor block compared with providing local anesthetic as a continuous basal infusion at an equivalent hourly dose.

DETAILED DESCRIPTION:
This investigation will be a randomized, observer-masked, controlled, split-body, human-subjects clinical trial. Of note, we will be using standard-of-care local anesthetics under their FDA approved purpose and do not plan to research a possible change of indication or use of these drugs as part of this research project.

Enrollment. Subjects will be volunteers of both sexes, age 18 and older. Volunteers will be solicited using newspaper advertisements, fliers, the CTRI Research Match, and an existing database of volunteers (IRB approved). If a volunteer meets inclusion/exclusion criteria and desires study participation, written, informed consent will be obtained. Selection for inclusion will not be based on race or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. A urine pregnancy test will be administered to all women of childbearing age following written informed consent but before any study interventions. This urine test will be administered by CTRI nursing staff using standard, FDA-approved urine pregnancy testing devices.

Inclusion and Exclusion Criteria. See section #10 below.

Perineural catheter insertion. Following written, informed consent, subjects will be admitted to the UCSD CTRI Center for Clinical Research Services (CCR) inpatient unit and have demographic/morphometric data recorded (e.g., age, weight, height). An intravenous line will be placed in an upper extremity, followed by external monitors (pulse oximeter, blood pressure, and EKG), and oxygen by nasal cannula. Sedation will be provided with intravenous fentanyl (50 μg) and/or midazolam (1 mg), or oral valium (10 mg) and/or dilaudid (4 mg), as necessary. Subjects will then have bilateral adductor canal perineural catheters placed using standard UC San Diego techniques.

Treatment Group Assignment. Subjects will act as their own controls: The dominant side (left or right) will be randomized to one of two treatment groups: ropivacaine 0.2% administration as either a basal infusion (8 mL/h) or bolus doses (8 mL administered hourly). The non-dominant contralateral side will receive the other possible treatment. Randomization will be based on computer-generated codes. Randomization will be in blocks of two, and stratified by sex. An infusion pump with study infusate will be attached to each of the perineural catheters and initiated at Hour 0. The basal rate and bolus volume will depend upon the treatment group (note that the basal rate and bolus volume differ for each treatment group, but the total dose of local anesthetic is the same for each):

Treatment Group Basal Rate (mL/h) Basal Dose (mg/h) Bolus Volume (mL) Bolus Dose (mg) Total Dose (mg/h) Basal Infusion 8 16 0 0 16 Bolus Doses 0 0 8 16 16

The tubing from the pumps to the subjects will be gently wound at least 5 rotations and covered with opaque tape, masking which perineural catheter is receiving which treatment (ropivacaine is clear, so the flow through the clear tubing from the tape to the perineural catheters will not be visually distinguishable).

Local Anesthetic Administration. The infusion pump administering the basal infusion will be initiated at Hour 0. The infusion pump administering bolus doses will administer a 8 mL bolus dose each hour beginning at Hour 0. Perineural catheters will be removed after 8 hours.

To check the perineural catheter placement accuracy, the adductor canal nerve block will be evaluated 8 hours after local anesthetic initiation and considered successful when subjects experience a decreased sensation to cold of the skin in the saphenous nerve distribution as compared with their ipsilateral upper extremity. Subjects will be deemed non-responders if both extremities failed to exhibit any increase in tolerance to cutaneous electrical current by Hour 8. For unsuccessful perineural catheter insertion, non-responders, or if a perineural catheter is inadvertently dislodged prior to the measurement of the primary endpoint, the data will not be included in the analyses and the subject dropped from the study.

Food and Drink: Both food and accompanying beverages/water will be provided by the hospital and served by the nursing staff immediately following catheter insertion. Meals will be provided without charge to the study subjects. There is no restriction on oral intake following catheter insertion. Subjects will remain within the CTRI-CCR until the following morning for the final measurement.

Outcome Measurements. We have selected measures that have established reliability and validity. Staff blinded to treatment group assignment will perform all measures and assessments. Measurements will be performed prior to local anesthetic administration initiation ("baseline"; Hour 0); as well as hourly following local anesthetic infusion/bolus initiation through Hour 14 (and one final measurement set prior to discharge the following morning at approximately Hour 22; see Table below). For all measurements, the dominant side will always be tested first, followed by the contralateral side.

Tolerance of transcutaneous electrical stimulation: Evaluated in the seated position using transcutaneous electrical stimulation (TES) in the same manner as described throughout the anesthesia literature (this is a "gold standard" for regional anesthesia studies). EKG pads will be positioned over the proximal patella and quadriceps tendon 1 cm medial of midline and attached to a nerve stimulator. The current will be increased from 0 mA until the subject reports slight discomfort (or, up to a maximum of 80 mA), at which time the current is recorded as the TES value and the nerve stimulator turned off.

Quadriceps femoris muscle strength: Evaluated using a portable isometric force dynamometer to measure the maximum voluntary isometric contraction (MVIC) in a seated position. The primary end point will be the quadriceps femoris maximum voluntary isometric contraction (MVIC) expressed as a percentage of the pre-ropivacaine (baseline) MVIC: post / pre x 100; with the two sides of each subject compared with each other at Hour 8.

Statistical Analysis Plan. We will assess the noninferiority of the bolus method (hourly 8 mL ropivacaine 0.2% bolus doses) compared to basal infusion (ropivacaine 0.2% 8 mL/h continuous basal infusion) on the primary endpoint of tolerance to cutaneous current at 8 hours using a 1-tailed t-test at the 0.025 significance level with an a priori-specified noninferiority delta of 10 mA. A value of 10 mA is determined a priori to be the smallest difference that would be clinically important between groups. This value is considered the minimally clinically-relevant current since it approximates the tolerated electrical current range at baseline of the general population-in other words, natural variability and therefore a relatively small amount of current to detect. A positive test for noninferiority will be accompanied by the 95% confidence interval (0.025 in the hypothesized direction) for the difference in means not including the noninferiority delta.

Secondary analysis will assess noninferiority of the bolus to the basal infusion method on mean tolerance to cutaneous current across all time points measured, using a noninferiority delta of 10 mA as above. In this repeated measures setting, noninferiority will be assessed in the context of a linear mixed model adjusting for the within-subject correlation (using an auto-regressive correlation structure). If the time-by-group interaction is non-significant (P>0.20) we will assess noninferiority collapsing over time and constructing a 1-tailed t-test (using noninferiority delta of 10 mA) based on the model-based treatment effect for bolus versus basal infusion. In presence of a group-time interaction noninferiority will be assessed separately at each time point and a Holm-Bonferroni correction made for multiple comparisons to maintain the hypothesis-wise type I error at 0.025.

We will also assess noninferiority of bolus to basal infusion on the secondary endpoint of quadriceps femoris MVIC (22 hours total) using a mixed effects model as described above.

The rejection region for a noninferiority test includes superiority, by definition (i.e., "not worse" implies either equivalent or better). Therefore, if bolus is found to not only be noninferior, but also superior, we will be able to claim superiority. This will be evidenced by the 95% CI for the difference between means falling above zero.

Although we hypothesize that the bolus method will be noninferior to basal infusion, it is possible that basal infusion would be noninferior to bolus. Therefore, we will also conduct the above tests assessing noninferiority of basal infusion to bolus. If noninferiority is found in both directions, we will claim equivalence at ±10mA. SAS software 9.3 (SAS Institute, Cary, NC, USA) and R software versions 2.15.3 (The R Foundation for Statistical Computing, Vienna, Austria) will be used for all analyses.

Sample Size Estimation. Sample size calculations are based on the primary aim of determining the relationship between perineural ropivacaine delivery technique (basal vs. bolus) and continuous adductor canal nerve block effects. To this end, we will perform a noninferiority trial with the primary endpoint designated as the maximum tolerance to transcutaneous electrical stimulation at Hour 8. With 24 subjects we will have approximately 90% power (88%) at the 0.025 significance level to detect noninferiority of bolus ropivacaine to basal infusion ropivacaine on mean tolerance to transcutaneous electrical stimulation at Hour 8 using an a priori noninferiority delta of 10 mA. Based on previously-published data, this conservatively assumes a standard deviation of tolerance difference between legs of 15 mA.

We will apply the same analysis of percent change from baseline at Hour 0 to the secondary outcome measures. We will also examine the time profiles of the responses over time with spaghetti and mean plots. Further secondary analyses will include mixed-effects modeling of the repeated hourly measures to confirm the analysis of percent change at 8 hours. These models will account for the hierarchical correlation of paired measures from each subject over time. We will use these models to test the effects of subject characteristics, including handedness, sex, height, weight, body mass index, and age.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥ 18 years; and (2) willing to have bilateral adductor canal perineural catheters placed with subsequent ropivacaine administration and motor/sensory testing for 14 hours, requiring an overnight stay in the UCSD CTRI-CCR to allow dissipation of local anesthetic infusion effects by the following morning.

Exclusion Criteria:

* (1) current daily analgesic use; (2) opioid use within the previous 4 weeks; (3) any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles; (4) morbid obesity [weight > 35 kg/m2]; (5) pregnancy (as determined by a urine pregnancy test prior to any study interventions); and (6) incarceration. We expect to recruit a maximum of 30 healthy volunteers; with a target goal of 24 for the analysis. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. There will be no participants from vulnerable populations, such as pregnant women, children, or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monahan AM, Sztain JF, Khatibi B, Furnish TJ, Jaeger P, Sessler DI, Mascha EJ, You J, Wen CH, Nakanote KA, Ilfeld BM. Continuous Adductor Canal Blocks: Does Varying Local Anesthetic Delivery Method (Automatic Repeated Bolus Doses Versus Continuous Basal Infusion) Influence Cutaneous Analgesia and Quadriceps Femoris Strength? A Randomized, Double-Masked, Controlled, Split-Body Volunteer Study. Anesth Analg. 2016 May;122(5):1681-8. doi: 10.1213/ANE.0000000000001182. PMID 26863502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a split-body study design, so while there were 24 human subjects involved; each had two treatments: one bolus and one basal. Therefore there were 24 sides receiving the "bolus" treatment and 24 sides receiving the "basal" treatment
Groups:
- Right Side Bolus, Left Side Basal: The right side received ropivacaine 0.2% administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses. Since it is a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as a continuous basal infusion (8 mL/h) for 8 hours total.
- Right Side Basal, Left Side Bolus: The right side received ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) for 8 hours total. Since it was a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses.
Period: Overall Study
Arm/Group | Right Side Bolus, Left Side Basal | Right Side Basal, Left Side Bolus
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Right Side BOLUS and Left Side BASAL: The right side received ropivacaine 0.2% administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses. Since it is a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as a continuous basal infusion (8 mL/h) for 8 hours total.
- Right Side BASAL and Left Side BOLUS: The right side received ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) for 8 hours total. Since it was a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses.
- Total: Total of all reporting groups
Arm/Group | Right Side BOLUS and Left Side BASAL | Right Side BASAL and Left Side BOLUS | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Height [Mean (Standard Deviation); unit: cm] | 173 (8) | 175 (10) | 174 (9)
Weight [Mean (Standard Deviation); unit: kg] | 74 (12) | 79 (14) | 76 (13)
Dominant Leg was the RIGHT leg [Number; unit: participants] — Just as with "handedness", people have a dominant lower extremity, or leg--it is usually the leg that people use to kick a ball.
  participants | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Tolerance to Cutaneous Electrical Current
Description: Evaluated in the seated position using transcutaneous electrical stimulation (TES) in the same manner as described throughout the anesthesia literature (this is a "gold standard" for regional anesthesia studies). EKG pads will be positioned over the proximal patella and quadriceps tendon 1 cm medial of midline and attached to a nerve stimulator. The current will be increased from 0 mA until the subject reports slight discomfort (or, up to a maximum of 80 mA), at which time the current is recorded as the TES value and the nerve stimulator turned off.
Time Frame: After 8 h of infusion
Measure: Mean (Standard Deviation); unit: mA
Groups:
- BOLUS: The right side received ropivacaine 0.2% administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses. Since it is a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as a continuous basal infusion (8 mL/h) for 8 hours total.
- BASAL: The right side received ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) for 8 hours total. Since it was a split body study, the left side of the body of these participants received ropivacaine 0.2% perineural administration as repeated 8 mL bolus doses starting at time point 0 and given hourly for 7 additional doses.
Arm/Group | BOLUS | BASAL
Number analyzed (Participants) | 24 | 24
mA | 26.6 (12.1) | 27.1 (14.5)

2. Secondary Outcome: Tolerance to Transcutaneous Electrical Current
Description: as for outcome 1
Time Frame: baseline through Hour 14 (except Hour 8 which is the primary outcome) and then again at Hour 22
Measure: Mean (Standard Deviation); unit: mA (milliamperes)
Groups:
- BOLUS: Bilateral adductor canal catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as hourly bolus doses of 8 mL each a total of 8 times: one at time point zero and 1 on the hour for the following 7 hours. For the left catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 8 hours
  Bolus: An adductor canal catheter was inserted and ropivacaine 0.2% administered as hourly bolus doses of 8 mL each: one at time point zero and then on the hour for 7 additional doses.
  Basal: An adductor canal catheter was inserted and ropivacaine 0.2% administered as a continuous basal infusion (8 mL/h) from time point zero for a total of 8 hours.
- BASAL: Bilateral adductor canal catheters were inserted and ropivacaine 0.2% administered concurrently. For the right catheter, the ropivacaine was administered as a continuous basal infusion (8 mL/h) from time point zero for the following 8 hours. For the left catheter, the ropivacaine was administered as hourly bolus doses of 8 mL each a total of 8 times: one at time point zero and 1 on the hour for the following 7 hours.
  Bolus: An adductor canal catheter was inserted and ropivacaine 0.2% administered as hourly bolus doses of 8 mL each: one at time point zero and then on the hour for 7 additional doses.
  Basal: An adductor canal catheter was inserted and ropivacaine 0.2% administered as a continuous basal infusion (8 mL/h) from time point zero for a total of 8 hours.
Arm/Group | BOLUS | BASAL
Number analyzed (Participants) | 24 | 24
mA (milliamperes)
  Baseline | 26.7 (7.6) | 26.6 (7.2)
  Hour 1 | 26.8 (8.8) | 24.7 (7.8)
  Hour 2 | 27.9 (9.0) | 27.4 (8.2)
  Hour 3 | 27.8 (9.6) | 29.7 (13.3)
  Hour 4 | 30.0 (14.0) | 29.7 (14.6)
  Hour 5 | 29.5 (13.7) | 30.1 (14.5)
  Hour 6 | 29.0 (14.0) | 29.0 (14.8)
  Hour 7 | 26.8 (12.1) | 25.9 (11.3)
  Hour 9 | 22.7 (8.8) | 24.3 (10.6)
  Hour 10 | 22.6 (8.6) | 24.9 (10.5)
  Hour 11 | 21.1 (8.4) | 25.0 (12.1)
  Hour 12 | 21.3 (7.8) | 24.6 (12.7)
  Hour 13 | 21.2 (7.4) | 23.2 (9.4)
  Hour 14 | 21.1 (7.9) | 22.3 (8.8)
  Hour 22 | 24.1 (8.8) | 24.5 (9.0)

3. Secondary Outcome: Maximum Voluntary Isometric Contraction of the Quadriceps
Description: Strength of the quadriceps muscle was assessed by measurement of maximum voluntary isometric contraction. In the sitting position, without using accessory muscle groups, subjects performed maximum forceful knee extension against an electromechanical dynamometer (MicroFET2, Lafayette Instrument Company, Lafeyette, IN). The subject sat at the side of the bed with their legs dangling. The device was placed against the anterior tibia just above the malleoli between the subject and a nonelastic 5 cm-wide fabric band that was affixed to the gurney to stabilize the dynamometer during flexing of the quadriceps femoris muscle. Subjects were instructed to come to maximum force of knee extension over 2 seconds, hold this force for 5 seconds, and then relax. The maximum force was recorded, and results are reported relative to the pre-infusion baseline measurement (i.e., percent of baseline).
Time Frame: Baseline and then every hour through Hour 14, as well as Hour 22
Measure: Mean (Standard Deviation); unit: percentage of baseline MVIC
Arm/Group | BOLUS | BASAL
Number analyzed (Participants) | 24 | 24
percentage of baseline MVIC
  Baseline | 188 (65) | 188 (78)
  Hour 1 | 84 (27) | 88 (36)
  Hour 2 | 89 (21) | 87 (30)
  Hour 3 | 95 (25) | 93 (32)
  Hour 4 | 92 (34) | 87 (31)
  Hour 5 | 95 (38) | 90 (29)
  Hour 6 | 88 (34) | 93 (91)
  Hour 7 | 85 (35) | 92 (29)
  Hour 8 | 88 (31) | 94 (32)
  Hour 9 | 86 (30) | 87 (30)
  Hour 10 | 89 (36) | 90 (32)
  Hour 11 | 89 (36) | 87 (30)
  Hour 12 | 87 (35) | 84 (29)
  Hour 13 | 84 (32) | 89 (31)
  Hour 14 | 85 (30) | 88 (29)
  Hour 22 | 114 (35) | 119 (39)

ADVERSE EVENTS:
Time Frame: 22 hours after intervention
Groups:
- Bolus: ropivacaine 0.2% administration as repeated, scheduled (one/h) bolus doses (8 mL) x8 h
  ropivacaine
- Basal: ropivacaine 0.2% administration as a continuous basal infusion (8 mL/h) x8 h
  ropivacaine
Arm/Group | Bolus | Basal
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No